CLINICAL TRIAL: NCT00405002
Title: A Validation Study of a New System for Measuring the End Expiratory Lung Volume During Mechanical Ventilation Acute in Intubated Patients
Brief Title: A Validation Study of a New System for Measuring the End Expiratory Lung Volume During Mechanical Ventilation
Status: Completed | Type: Observational
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Davide Chiumello, MD, Policlinico Hospital
Other Study IDs: 101020
Record Dates: First submitted 2006-11-27; First posted 2006-11-29 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Respiratory Failure
Keywords: Acute respiratory failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: ALI/ARDS patients
  Interventions: Procedure: Helium dilution technique, lung CT scan

INTERVENTIONS:
Procedure: Helium dilution technique, lung CT scan — Helium dilution technique and lung CT scan

SUMMARY:
In this study the investigators aim to evaluate a new system dedicated to estimate the end expiratory lung volume, by measuring the VO2-VCO2, during mechanical ventilation compared to the helium dilution technique and the computed tomography (CT) scan.

DETAILED DESCRIPTION:
In this study we aimed to evaluate a new system dedicated to estimate the end expiratory lung volume, by measuring the VO2-VCO2, during mechanical ventilation compared to the Helium dilution technique and the CT scan. We will compare the data considering the CT scan data as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Adult intubated subjects

Exclusion Criteria:

* Barotrauma

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ALI/ARDS patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2006-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davide Chiumello, MD, Principal Investigator — Policlinico Hospital
Locations (1):
- Policlinico Hospital, Milan, Italy

REFERENCES:
- [Derived] Chiumello D, Cressoni M, Chierichetti M, Tallarini F, Botticelli M, Berto V, Mietto C, Gattinoni L. Nitrogen washout/washin, helium dilution and computed tomography in the assessment of end expiratory lung volume. Crit Care. 2008;12(6):R150. doi: 10.1186/cc7139. Epub 2008 Dec 1. PMID 19046447